CLINICAL TRIAL: NCT00739310
Title: A Pilot Study to Assess the Efficacy and Effectiveness of High-Frequency Chest Wall Oscillation (HFCWO) in Preventing Pulmonary Exacerbations in Children With Muscle Weakness and Restrictive Lung Disease CR-0088
Brief Title: Study Assessing High-Frequency Chest Wall Oscillation (HFCWO) in Preventing Pulmonary Exacerbations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hill-Rom (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CR-0088
Record Dates: First submitted 2008-08-20; First posted 2008-08-21 (Estimated); Results first posted 2015-09-24 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-07

CONDITIONS: Cerebral Palsy
Keywords: High Frequency Chest Wall Oscillation; Cerebral Palsy; Restrictive lung disease
MeSH Terms: conditions — Cerebral Palsy | interventions — Chest Wall Oscillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vest Treatment (HFCWO) (Experimental): Patients will receive Vest treatments for airway clearance therapy 2 x daily for 12 months. These data will be compared to 12 months of data prior to Vest initiation.
  Interventions: Device: Vest Treatment (high frequency chest wall oscillation)

INTERVENTIONS:
Device: Vest Treatment (high frequency chest wall oscillation) — twice daily for 15-20 minutes
  Other Names: HFCWO

SUMMARY:
To asssess efficacy of airway clearance provided by Vest therapy (HFCWO) in the reduction of respiratory exacerbations requiring hospitalization or antibiotic utilization in patients with muscle weakness and restrictive lung disease.

DETAILED DESCRIPTION:
This non-randomized home based pre-post intervention study. The study will compare the efficacy of Vest® therapy (HFCWO) for mucus secretion clearance in a population of patients with muscle weakness and restrictive lung disease with frequent pulmonary exacerbations. Enrolled subjects with a tracheostomy will be evaluated for microbial load and inflammatory status as a pilot evaluation of microbial load and inflammatory status outcomes.

The total number of evaluable subjects to be recruited is estimated at 40. Subjects will be considered evaluable if they have completed at least 6 months of follow up.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 months old.
* Subject has a chest circumference of greater than 19 inches.
* Subject has a diagnosis of muscle weakness and restrictive lung disease.
* Ability to provide Informed consent from legal guardian.
* Subject has had 2 or more exacerbations requiring either hospitalization or antibiotics (IV or oral) in the past 12 months
* If inhaled Tobramycin has been prescribed prophylacticly, subjects must discontinue the medication at least 2 weeks prior to study enrollment

Exclusion Criteria:

* Subject has a diagnosed allergy with a respiratory trigger.
* Participation in another clinical trial.
* Unstable head or spinal injury.
* Unresolved pneumothorax or pneumomediastinum present
* Unresolved hemorrhage
* Hypotension requiring vasopressors or positioning
* Bronchopleural fistula
* Gross hemoptysis within the past eight hours
* Pulmonary embolism or history of pulmonary embolism within the past two months
* Burns, open wounds and skin infections on the thorax
* Osteomyelitis of the ribs
* Osteoporosis with history of fractures.

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2008-08; Primary Completion 2010-10 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikail Kazachkov, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vest Treatment (HFCWO): Patients will receive Vest treatments for airway clearance therapy 2 x daily
  Vest Treatment (high frequency chest wall oscillation): twice daily for 15-20 minutes
Period: Overall Study
Arm/Group | Vest Treatment (HFCWO)
Started | 29
Completed | 22
Not Completed | 7
Not completed — Poor adherance to prescribed therapy | 4
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Patients who completed 12 months of prospective therapy
Arm/Group | Vest Treatment (HFCWO)
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.55 (5.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Hospitalizations Lasting at Least 24 Hours in This Patient Population
Description: Hospitalizations lasting at least 24 hours
Time Frame: end of study
Measure: Number; unit: hospitalizations
Groups:
- Pre-Treatment: Prior to Vest Treatment
- Post Vest Treatment: 12 months of intervention 2 x daily Vest Therapy
Arm/Group | Pre-Treatment | Post Vest Treatment
Number analyzed (Participants) | 22 | 22
hospitalizations | 10 | 8

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Vest Treatment (HFCWO)
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

LIMITATIONS AND CAVEATS:
Study design was sub-optimal due to lack of control group and lack of randomization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No